CLINICAL TRIAL: NCT02081469
Title: Phase IV; Different Extend Treatment Duration (6 Months vs 12 Months After Chemotherapy) to Prevent HBV Relapse With Tenofovir for Prophylaxis in Patients With Malignant Tumor Combined With HBV Carrier Receiving Chemotherapy
Brief Title: Prophylaxis of CHB Patients With Malignant Tumor Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Chao-Wei Hsu, MD, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: IN-US-174-0207
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis B, Chronic; Tumor
Keywords: Chronic hepatitis B; HBV; Chemotherapy; Reactivation; Prophylaxis
MeSH Terms: conditions — Hepatitis B, Chronic; Neoplasms | interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: Tenofovir 300mg QD. Two arm: 6 month and 12 month.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A:TDF for extend 24 weeks (Other): Arm A:Continue TDF 300mg daily for extend 24 weeks after completion of chemotherapy
  Interventions: Other: TDF
- Arm B: TDF for extend 48 weeks (Other): Arm B: Continue TDF 300mg daily for extend 48 weeks after completion of chemotherapy.
  Interventions: Other: TDF

INTERVENTIONS:
Other: TDF — To compare extend TDF 24 wks versus 48 wks prophylaxis efficacy in chemotherapy CHB patients
  Other Names: viread

SUMMARY:
To evaluate the effectiveness and safety of tenofovir for different treatment duration in preventing HBV relapse in patients with malignancies after receiving chemotherapy and off-treatment of chemotherapy.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness and safety of tenofovir in preventing HBV relapse in HBV carriers with malignant tumor following chemotherapy. Approximately 100 patients who are planned to receive chemotherapy for malignant tumor will be invited to participate in this trail. A 1 or less 1-week tenofovir prophylaxis treatment should be administered by all subjects prior to the chemotherapy and eligible subjects will be randomly assigned to extend 24-week prophylaxis group A or 48-week prophylaxis group B in a 1:1 ratio at the end of the chemotherapy. The subjects could be stopped or withdrawn from this study earlier if HBV relapses or need to receive another course of chemotherapy respectively. The relapse episode will be followed until 24 weeks after the end of prophylaxis therapy. Data collection will take place at screening, every cyclic visit of chemotherapy, at the end of chemotherapy, and the following prophylaxis period, then every 4 weeks during the follow-up period. Patients in both groups will be treated with tenofovir or other antiviral agent according to investigator judgement when HBV relapse after discontinuation of tenofovir therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 70 years of age
2. Patients with histologically proven malignant tumor planned to receive chemotherapy after enrollment
3. Hepatitis B virus (HBV) carriers who fulfill one of the following criteria:

   seropositive of HBsAg, or HBsAg negative, but Anti-HBc positive with HBV DNA detectable defined as HBV DNA > 20 IU/mL (by Roche Taqman real time assay).
4. Patients with ALT ≤ 2 x ULN (upper limit of normal)
5. Normal Cr mg/dL or eGFR > 80 mL/min
6. Life expectancy > 1 year
7. Willing and able to provide written informed consent

Exclusion Criteria:

1. Females who are pregnant/nursing or with intention to be pregnant within the study period
2. Documented hepatitis C virus (HCV) co-infection
3. Patients with other current major systemic disease such as active infection, significant cardiac disease, poor control diabetes mellitus, osteopenia or osteoporosis that the investigators consider to be significant risk
4. Current use of any hepatitis B prophylaxis medication
5. Decompensated liver cirrhosis
6. Current or previous use of any chemotherapy
7. Use of any investigational product medicine within 1 month prior to the initiation of study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
To compare the HBV relapse rate during the follow-up period in HBV carriers with malignant tumor receiving tenofovir for 24 and 48 weeks after the end of chemotherapy. | 24 to 48 weeks
  To compare the HBV relapse rate during the follow-up period in HBV carriers with malignant tumor receiving tenofovir for 24 and 48 weeks after the end of chemotherapy.
  * HBV relapse is defined as: acute liver flare, i.e. ALT ≥ 2 x ULN and HBV DNA > 2000 IU/mL.

SECONDARY OUTCOMES:
To estimate the efficacy of TDF during chemotherapy with after chemotherapy and post-chemotherapy,as measure by the HBV reactivation, clinical relapse and adverse events in all patients. | The efficacy of TDF duration 24 wks versus 48 wks extended
  AST, ALT, Bil(T), Cr (eGFR or MDRD), phosphate, urine analysis, HBsAgQT and HBV DNA were measured at baseline, every 2 cycle of chemotherapy, the end of chemotherapy, the end of TDF and the end of complete follow-up (after the end of TDF for 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Wei Hsu, MD, Principal Investigator — Chang Gung Medical Foundation (Linkou Branch)
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu CW, Chen SC, Wang PN, Wang HM, Chen YC, Yeh CT. Preventing viral relapse with prophylactic tenofovir in hepatitis B carriers receiving chemotherapy: a phase IV randomized study in Taiwan. Hepatol Int. 2024 Apr;18(2):449-460. doi: 10.1007/s12072-023-10635-5. Epub 2024 Feb 20. PMID 38376651